CLINICAL TRIAL: NCT03334357
Title: Physical Fitness as Klotho Protein Stimulator; Antiaging Effects of New Training Methods (FIT-AGING).
Brief Title: Physical Fitness as Klotho Protein Stimulator.
Acronym: FIT-AGING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuel Castillo Garzón (Other)
Responsible Party: Sponsor-Investigator, Manuel Castillo Garzón, University professor, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FPU14/04172
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Physical Activity; Aging
Keywords: Physical fitness; Klotho; Training; HIIT; WB-EMS
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Non-Exercise group. We will provide general advices to control group participants thought an information meeting performed by a graduate in Sport Sciences. It will recommended to follow the physical activity recommendations for adults provided by World Health Organization
- PAR group (Experimental): The volume in PAR is based on the minimum physical activity recommended (150min/week at moderate intensity).
  Intensity selected for PAR aerobic training is 60-65% HRres. Strength intensity selected was 40-50% of 1 RM.
  Frequency. PAR group will train 3 days/week, the minimum frequency recommended. Exercises programmed for the aerobic exercise are treadmill, cycle-ergometer and elliptical ergometer in aerobic training part and weight bearing and guided pneumatic machines (involved major upper and lower body muscle group) in resistance training.
  Training load variation. We propose a gradual progression to control the exercise dose Training periodization divided in two phases of 5 weeks each one, starting with a familiarization phase (2 weeks).
  Training sessions. Sessions start with a dynamic standardized warm up, which include several muscle activation exercises. Aerobic sessions include compensatory exercises. Training session will be ended with a cooling-down protocol
  Interventions: Other: PAR
- HIIT group. (Experimental): The volume in HIIT 40-65 min/week at high intensity. Intensity. Two different protocols: HIIT with long intervals (Type A session), which intensity will be >95% VO2max and HIIT with short intervals (Type B session), >120% VO2max.
  Training frequency two times/week. Type of exercise. Type A session are walking in treadmill with personalized slopes. Eight weight-bearing exercises in circuit form, type B session.
  Training load variation. Gradual progression to control the exercise dose. Training periodization divided in: familiarization phase, phase I, phase II. Training sessions. Type A: 5 minutes in treadmill at 60% VO2max. After warm-up, participants complete sets corresponding to each training session following the corresponding characteristics. Type B: eight weight-bearing exercises (in circuit form) two times/set with an active rest (walking at 60%VO2max) as many times at as defined. Training session will be ended with a cooling-down protocol
  Interventions: Other: HIIT
- WB-EMS group. (Experimental): WB-EMS training program will be the same than HIIT intervention related to volume, intensity, frequency, type of exercise, training load variation, training periodization and training session. However, electrical impulse will be included in order to assess if WB-EMS training will produce an added effect compared to HIIT.
  Electrical parameters:
  We will apply a frequency of 15-33 Hz in type A session. And, we will apply a frequency of 35-75 Hz in type B session.
  Intensity will be 80-100 mA. Impulse Width adjusted in relation to body segment: thigh zone (400μsec), glute zone (350μsec), abdominal zone (300μsec), dorsal zone (250μsec), cervical (200μsec), chest zone (200μsec) and arm zone (200μsec).
  Duty cycle. We have programmed a duty cycle of 50-67% in type B session, but duty cycle in type A session will be 99%.
  RPE impulse: the impulse intensity was individually adapted to generate similar values of rate of perceived exertion (RPE) in Borg CR-10 Scale "5" of "9"
  Interventions: Other: WB-EMS

INTERVENTIONS:
Other: PAR
  Arms: PAR group
Other: HIIT
  Arms: HIIT group.
Other: WB-EMS
  Arms: WB-EMS group.

SUMMARY:
FIT-AGING will determine the effect of different exercise modalities on α-Klotho protein (primary outcome) in sedentary healthy adults. FIT-AGING also investigate the physiological consequences of activating Klotho gene (secondary outcomes).

DETAILED DESCRIPTION:
Aims: The plasma Klotho protein concentration (α-Klotho protein), which is considered a powerful biomarker of longevity, makes it an attractive target as an anti-aging therapy against functional decline, sarcopenic obesity, metabolic and cardiovascular diseases, osteoporosis, and neurodegenerative disorders. Physical exercise and physical fitness, could be α-Klotho protein activators through biochemical process. FIT-AGING will determine the effect of different exercise modalities on α-Klotho protein (primary outcome) in sedentary healthy adults. FIT-AGING also investigate the physiological consequences of activating Klotho gene (secondary outcomes).

Methods: FIT-AGING will recruit 60 sedentary, healthy, adults (50% women) aged 40-65 years. Eligible participants will be randomly assigned to a non-exercise group to the usual control group (n=15), physical activity recommendation from American College of Sport Medicine, World Health Organization and American Heart Association group (n=15), High Intensity Interval Training group (n=15)) and Whole-Body Electromyostimulation group (n=15). Laboratory measures completed at baseline and 12 weeks later, include α-Klotho protein concentration, physical fitness (cardiorespiratory fitness, muscular strength), body composition, resting metabolic rate, hearth rate variability (HRV), health blood biomarkers, free-living physical activity, sleep habits reaction time, cognitive variables and health-related questionnaires. The investigators will also obtain dietary habits data and cardiovascular disease risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-65 years
* BMI:18.5-35 kg/m2
* Not engaged in regular physical activity >20min on >3days/week
* Not participating in a weight loss programme
* Stable weight over the last 5 months (body weight changes>5kg)
* Participant must be capable and willing to provide consent, understand exclusion criteria and accept the randomized group assignment
* Normal electrocardiogram

Exclusion Criteria:

* History of cardiovascular disease
* Diabetes
* Pregnancy or planning to get pregnant during study period
* Beta blockers or benzodiapezins use
* Taking medication for thyroid
* Other significant conditions that are life-threatening or that can interfere with or be aggravated by exercise
* Unwillingness to either complete the study requirements or to be randomized into control or training group
* A first-degree relative with history of cancer

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2017-12-23 (Actual)

PRIMARY OUTCOMES:
α-Klotho protein | Baseline and through study completion, an average of 12 weeks.
  Plasma Klotho concentrations will be measured by ELISA using a soluble α-Klotho ELISA assay kit.

SECONDARY OUTCOMES:
Physical fitness: cardiorespiratory fitness | Baseline and through study completion, an average of 12 weeks.
  Cardiorespiratory fitness measure through a maximum treadmill test (VO2max.).
Physical fitness: muscular strength. | Baseline and post-intervention.Baseline and through study completion, an average of 12 weeks.
  Muscle strength measure through: Isokinetic strength, Handgrip strength and Core resistance stability.
Body composition. | Baseline and through study completion, an average of 12 weeks.
  Measure by DXA.
Resting energy expenditure. | Baseline and through study completion, an average of 12 weeks.
  Evaluated by indirect calorimetry with gas analyzer breath by breath.
Hearth Rate Variability (HRV). | Baseline and through study completion, an average of 12 weeks.
  Measure by Polar RS800CX.
Biochemical profile. | Baseline and through study completion, an average of 12 weeks.
  General biochemical profile in blood samples
Physical activity. | Baseline and through study completion, an average of 12 weeks.
  The amount of physical activity will be measured by accelerometer.
Reaction time. | Baseline and through study completion, an average of 12 weeks.
  Measure by Vienna System.
Cognitive test. | Baseline and through study completion, an average of 12 weeks.
  Auditory memory tests
Dietary assessment. | Baseline and post-Baseline and through study completion, an average of 12 weeks..
  Measure by 24h recall and Food Frecuency Questionnaire.
Anthopometric measures. | Baseline and post-Baseline and through study completion, an average of 12 weeks..
  Measure by stadiometer and scale.
Sleep quality. | Baseline and post-Baseline and through study completion, an average of 12 weeks..
  The quality of sleep will be measured by accelerometer.
Hormones profile | Baseline and post-Baseline and through study completion, an average of 12 weeks..
  Hormones profile measure in blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel J Castillo Garzón, Professor, Principal Investigator — Universidad de Granada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Navarro-Lomas G, Dote-Montero M, Alcantara JMA, Plaza-Florido A, Castillo MJ, Amaro-Gahete FJ. Different exercise training modalities similarly improve heart rate variability in sedentary middle-aged adults: the FIT-AGEING randomized controlled trial. Eur J Appl Physiol. 2022 Aug;122(8):1863-1874. doi: 10.1007/s00421-022-04957-9. Epub 2022 May 10. PMID 35538242
- [Derived] Dote-Montero M, De-la-O A, Jurado-Fasoli L, Ruiz JR, Castillo MJ, Amaro-Gahete FJ. The effects of three types of exercise training on steroid hormones in physically inactive middle-aged adults: a randomized controlled trial. Eur J Appl Physiol. 2021 Aug;121(8):2193-2206. doi: 10.1007/s00421-021-04692-7. Epub 2021 Apr 22. PMID 33890158
- [Derived] Jurado-Fasoli L, Amaro-Gahete FJ, Merchan-Ramirez E, Labayen I, Ruiz JR. Relationships between diet and basal fat oxidation and maximal fat oxidation during exercise in sedentary adults. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1087-1101. doi: 10.1016/j.numecd.2020.11.021. Epub 2020 Dec 1. PMID 33549436
- [Derived] De-la-O A, Jurado-Fasoli L, Castillo MJ, Gutierrez A, Amaro-Gahete FJ. 1,25-Dihydroxyvitamin D and S-Klotho Plasma Levels: The Relationship Between Two Renal Antiaging Biomarkers Mediated by Bone Mineral Density in Middle-Aged Sedentary Adults. Rejuvenation Res. 2021 Jun;24(3):227-233. doi: 10.1089/rej.2020.2384. Epub 2021 Mar 5. PMID 33487127
- [Derived] Amaro-Gahete FJ, Sanchez-Delgado G, Ara I, R Ruiz J. Cardiorespiratory Fitness May Influence Metabolic Inflexibility During Exercise in Obese Persons. J Clin Endocrinol Metab. 2019 Dec 1;104(12):5780-5790. doi: 10.1210/jc.2019-01225. PMID 31322652
- [Derived] Jurado-Fasoli L, Amaro-Gahete FJ, De-la-O A, Castillo MJ. Impact of different exercise training modalities on energy and nutrient intake and food consumption in sedentary middle-aged adults: a randomised controlled trial. J Hum Nutr Diet. 2020 Feb;33(1):86-97. doi: 10.1111/jhn.12673. Epub 2019 Jul 3. PMID 31270896